CLINICAL TRIAL: NCT00273962
Title: A Comparison of Combivent® UDV (Ipratropium 500mcg and Salbutamol 2.5mg) and Salbutamol UDV Alone (2.5mg) in a Double-Blind Efficacy and Safety Study in Asthmatic Children With Severe Acute Exacerbation
Brief Title: A Comparison of Combivent UDV (Ipratropium 500mcg and Salbutamol 2.5mg) and Salbutamol UDV Alone (2.5mg)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.45
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Ipratropium

INTERVENTIONS:
Drug: ipratropium plus salbutamol UDV
Drug: salbutamol UDV

SUMMARY:
To compare the bronchodilator efficacy of ipratropium plus salbutamol (Combivent) with salbutamol alone given every 20 minutes for three doses in asthmatic children with severe acute exacerbation

DETAILED DESCRIPTION:
A Comparison of Ipratropium 500mcg and salbutamol 2.5mg (Combivent UDV) and salbutamol UDV alone (2.5mg) in a Double-blind, Efficacy and Safety Study in Asthmatic Children with Severe Acute Exacerbation

Study Hypothesis:

Several studies, including a study conducted in an emergency room setting, demonstrated that the addition of ipratropium bromide, an anticholinergic drug, to standard salbutamol therapy significantly improves pulmonary function as compared to salbutamol alone.

Comparison(s):

Ipratropium bromide 500 mcg plus salbutamol 2.5mg (Combivent) vs salbutamol (2.5mg) alone given every 20 minutes for 3 doses

ELIGIBILITY:
INCLUSION CRITERIA

1. All patients must have a known history of asthma and present to the hospital/clinic with severe acute exacerbation.
2. Male or female patients 2 to 10 years of age.
3. Parents or legal guardians of patients must sign an Informed Consent Form prior to participation in the trial.

EXCLUSION CRITERIA

1. Patients with known or suspected hypersensitivity to study drugs
2. Patients with medical condition that would contraindicate the use of beta2-adrenergic or anticholinergic medications
3. Patients with first wheezing episode only
4. Prior intubation for asthma for more than 24 hours
5. Patients who used ipratropium within six hours prior to consultation
6. Patients with concurrent stridor or possible presence of intra-thoracic foreign body
7. Patients with disease known to have chronic effect on respiratory function ( e.g., cystic fibrosis or cardiac disease)
8. Patients requiring immediate resuscitation or airway intervention
9. With psychiatric disease or psychosocial problems
10. Patients on other investigational drugs or have used any other investigational drugs within the past month

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2002-05; Primary Completion 2003-11 (Actual); Study Completion 2003-11

PRIMARY OUTCOMES:
The proportion of patients showing improvement in asthma severity scores from severe at baseline to mild at the end of the treatment

SECONDARY OUTCOMES:
Change in asthma severity scores from baseline to end of treatment; number of patients needing hospitalization; number of rescue medications; oxygen saturation, number of discharged patients revisiting the ER/doctors clinic

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. (Phil) Inc.
Locations (10):
- Philippines (10):
  - Jose Reyes Memorial Medical Center, Manila
  - Philippine General Hospital, Manila
  - Amang Rodriguez Hospital, Marikina City
  - San Juan de Dios Hospital, Pasay
  - Rizal Provincial Hospital, Pasig
  - Philippine Children's Medical Center, Quezon
  - Quezon City General Hospital, Quezon
  - East Ave Medical Center, Quezon City
  - Philipines Heart Center, Quezon City
  - Quirino Memorial Medical Center, Quezon City